CLINICAL TRIAL: NCT04991753
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled, Proof-of-concept Study Evaluating the Efficacy and Safety of Nipocalimab Administered Intravenously in Participants With Active Rheumatoid Arthritis Despite Standard Therapy
Brief Title: A Proof-of-concept Study of the Efficacy and Safety of Nipocalimab in Participants With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109058; 80202135ARA2001 (Other: Janssen Research & Development, LLC); 2021-000510-42 (EudraCT Number)
Expanded Access: NCT05221619 (Temporarily not available)
Record Dates: First submitted 2021-08-02; First posted 2021-08-05 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Placebo (Placebo Comparator): Participants will receive placebo intravenously (IV) every 2 weeks (q2w) through Week 10 along with standard-of-care background therapy.
  Interventions: Other: Placebo
- Group 2: Nipocalimab (Experimental): Participants will receive nipocalimab IV q2w through Week 10 along with standard-of-care background therapy.
  Interventions: Drug: Nipocalimab

INTERVENTIONS:
Other: Placebo — Placebo infusion will be administered intravenously.
  Arms: Group 1: Placebo
Drug: Nipocalimab — Nipocalimab infusions will be administered intravenously.
  Other Names: JNJ-80202135; M281
  Arms: Group 2: Nipocalimab

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of nipocalimab versus placebo in participants with moderate to severe active rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
RA is a chronic autoimmune inflammatory disorder of unknown etiology that occurs in approximately 1 percent (%) of the population. Nipocalimab (also referred to as JNJ-80202135 and M281) is a fully human aglycosylated immunoglobulin (Ig)G1 monoclonal antibody designed to selectively bind, saturate, and block the IgG binding site on the endogenous neonatal fragment crystallizable (Fc) receptor (FcRn). Nipocalimab has a unique mechanism of action whereby it blocks the IgG binding site on endogenous FcRn and is expected to decrease pathogenic IgG antibody concentrations. A significant involvement of pathogenic IgG antibodies has been demonstrated in autoimmune diseases including RA. The primary hypothesis is that treatment with nipocalimab intravenously (IV) every 2 weeks (q2w) is superior to placebo in participants with moderate to severe active rheumatoid arthritis (RA) as assessed by the mean change from baseline in the disease activity index score 28 using C-reactive Protein (DAS28-CRP) at Week 12. The study consists of a Screening Period (less than or equal to [<=] 6 Weeks), Double-blind Treatment Period (12 Weeks), and a Safety Follow-up Period (6 Weeks). Key safety assessments will include adverse events (AEs), serious adverse events (SAEs), adverse events of special interests (AESIs), clinical laboratory safety tests (hematology, chemistry, and lipid profile), vital signs, and physical examination. The total duration of the study is up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis (RA) and meeting the 2010 American college of rheumatology (ACR)/European League Against Rheumatism (EULAR) criteria for RA for at least 3 months before screening
* Has moderate to severe active RA as defined by persistent disease activity with at least 6 swollen and 6 tender joints out of the 66/68-swollen and tender joint count at the time of screening and at baseline
* Is positive for anti-citrullinated protein antibodies (ACPA) and/or rheumatoid factor (RF) at screening
* Screening C-reactive protein (CRP) greater than or equal to (>=) 0.3 milligram per deciliter (mg/dL) by the central laboratory
* A woman of childbearing potential must have a negative highly sensitive urine pregnancy test (beta-human chorionic gonadotropin [beta-hCG]) at screening and a negative urine (beta-hCG) pregnancy test at Week 0 prior to administration of study intervention

Exclusion Criteria:

* Has any confirmed or suspected clinical immunodeficiency syndrome not related to treatment of his/her RA or has a family history of congenital or hereditary immunodeficiency unless confirmed absent in the participant
* Currently has a malignancy or has a history of malignancy within 3 years before screening (with the exception of localized basal cell carcinoma and/or squamous cell carcinoma skin cancer that has been adequately treated with no evidence of recurrence for at least 12 weeks before the first administration of study intervention or cervical carcinoma in situ that has been treated with no evidence of recurrence for at least 3 months before the first administration of study intervention)
* Is (anatomically or functionally) asplenic
* Has experienced myocardial infarction (MI), unstable ischemic heart disease, or stroke within 12 weeks of screening
* Has other known inflammatory diseases that might confound the evaluations of benefit from nipocalimab therapy, including but not limited to ankylosing spondylitis, psoriatic arthritis, systemic lupus erythematosus, Lyme disease
* Is currently taking immunoglobulin (Ig)G fragment crystallizable (Fc)-related protein therapeutics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (28):
- United States (13):
  - Arizona Arthritis & Rheumatology Associates PC, Glendale, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Mesa, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Tucson, Arizona
  - Desert Medical Advances, Palm Desert, California
  - Arthritis Care and Research Center Inc.: Smitha Reddy, MD, Poway, California
  - TriWest Research Associates, LLC, San Diego, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - STAT Research, Inc., Vandalia, Ohio
  - Low Country Rheumatology PA, Summerville, South Carolina
  - West Tennessee Research Institute, Jackson, Tennessee
  - Accurate Clinical Research, Inc., Houston, Texas
  - Southwest Rheumatology Research LLC, Mesquite, Texas
- Germany (2):
  - Hamburger Rheuma Forschungszentrum II, Hamburg
  - Rheumazentrum Ratingen, Ratingen
- Poland (4):
  - Szpital Uniwersytecki nr 2 im dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - NZOZ Lecznica Mak-Med sc, Nadarzyn
  - Prywatna Praktyka Lekarska Prof Um Dr Hab Med Pawel Hrycaj, Poznan
  - Centrum Medyczne AMED Targowek, Warsaw
- Spain (5):
  - Hosp Univ A Coruna, A Coruña
  - Hosp. Univ. de Basurto, Bilbao
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Virgen Macarena, Seville
  - Hosp. Do Meixoeiro, Vigo
- United Kingdom (4):
  - Western General Hospital, Edinburgh
  - Kings College Hospital NHS Trust, London
  - North Tyneside General Hospital, Newcastle
  - Haywood Hospital, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Taylor PC, Schett G, Huizinga TW, Wang Q, Ibrahim F, Zhou B, Liva SG, Shaik JSB, Xiong Y, Leu JH, Panchakshari RA, Loza MJ, Ma K, Dhatt H, Rojo Cella R, Karyekar CS, Cuff CA, Gao S, Fei K. Nipocalimab, an anti-FcRn monoclonal antibody, in participants with moderate to severe active rheumatoid arthritis and inadequate response or intolerance to anti-TNF therapy: results from the phase 2a IRIS-RA study. RMD Open. 2024 Jun 28;10(2):e004278. doi: 10.1136/rmdopen-2024-004278. PMID 38942592

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Placebo: Participants received placebo matched to nipocalimab as intravenous (IV) infusion every 2 weeks (q2w) from Week 0 through Week 10 along with standard-of-care background therapy. Participants were followed up for safety up to 8 weeks after administration of last study intervention at Week 10.
- Group 2: Nipocalimab: Participants received nipocalimab 15 milligrams per kilogram (mg/kg) as IV infusion q2w from Week 0 through Week 10 along with standard-of-care background therapy. Participants were followed up for safety up to 8 weeks after administration of last study intervention at Week 10.
Period: Overall Study
Arm/Group | Group 1: Placebo | Group 2: Nipocalimab
Started | 20 | 33
Completed | 20 | 32
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Placebo | Group 2: Nipocalimab | Total
Number analyzed (Participants) | 20 | 33 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (8.57) | 56.0 (12.30) | 56.9 (11.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 24 | 36
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 16 | 29 | 45
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 18 | 30 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Index Score 28 Using C-reactive Protein (DAS28-CRP) at Week 12
Description: Change from baseline in DAS28-CRP at Week 12 were reported. The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity, and C-reactive protein (CRP; in milligrams per liter [mg/L]). The set of 28 joint count was based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. Score on the DAS28 ranged from 0 to 10, where higher scores indicated more disease activity. Negative changes from baseline indicated improvement of arthritis.
Time Frame: Baseline (Week 0), Week 12
Population: The full analysis set (FAS) included all randomized participants who received at least 1 dose (partial or complete) of any study intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Group 1: Placebo | Group 2: Nipocalimab
Number analyzed (Participants) | 20 | 33
Score on a scale | -0.58 [-1.24 to 0.07] | -1.03 [-1.66 to -0.40]
Statistical Analysis 1: Comparison: Group 1: Placebo vs Group 2: Nipocalimab; Test type: Superiority; p = 0.224, ANCOVA; Least square mean difference = -0.45, 95% CI 2-sided [-1.17 to 0.28]

2. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology (ACR) 20 at Week 12
Description: Percentage of participants who achieved ACR20 at Week 12 were reported. ACR20 response is defined as: greater than or equal to (>=)20% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=20% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using visual analog scale (VAS; 0-100 millimeters [mm], 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function as measured by Disability Index of Health Assessment Questionnaire (HAQ-DI; 20-question instrument assessing 8 functional areas; range: 0-3, 0= no difficulty, 3= inability to perform task in that area), and CRP.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Placebo | Group 2: Nipocalimab
Number analyzed (Participants) | 20 | 33
Percentage of Participants | 20.0 [-1.24 to 0.07] | 45.5 [-1.66 to -0.40]

3. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology (ACR) 50 at Week 12
Description: Percentage of participants who achieved ACR50 at Week 12 were reported. ACR50 response is defined as: >=50% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=50% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using visual analog scale (VAS; 0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function as measured by Disability Index of Health Assessment Questionnaire (HAQ-DI; 20-question instrument assessing 8 functional areas; range: 0-3, 0= no difficulty, 3= inability to perform task in that area), and CRP.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Placebo | Group 2: Nipocalimab
Number analyzed (Participants) | 20 | 33
Percentage of Participants | 5.0 [-1.24 to 0.07] | 15.2 [-1.66 to -0.40]

4. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology (ACR) 70 at Week 12
Description: Percentage of participants who achieved ACR70 at Week 12 were reported. ACR70 response is defined as: >=70% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=70% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using visual analog scale (VAS; 0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function as measured by Disability Index of Health Assessment Questionnaire (HAQ-DI; 20-question instrument assessing 8 functional areas; range: 0-3, 0= no difficulty, 3= inability to perform task in that area), and CRP.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Placebo | Group 2: Nipocalimab
Number analyzed (Participants) | 20 | 33
Percentage of Participants | 0 [-1.24 to 0.07] | 12.1 [-1.66 to -0.40]

5. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology (ACR) 90 at Week 12
Description: Percentage of participants who achieved ACR90 at Week 12 were reported. ACR90 response is defined as: >=90% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=90% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using visual analog scale (VAS; 0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function as measured by Disability Index of Health Assessment Questionnaire (HAQ-DI; 20-question instrument assessing 8 functional areas; range: 0-3, 0= no difficulty, 3= inability to perform task in that area), and CRP.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Placebo | Group 2: Nipocalimab
Number analyzed (Participants) | 20 | 33
Percentage of Participants | 0 [-1.24 to 0.07] | 6.1 [-1.66 to -0.40]

6. Secondary Outcome: Percentage of Participants Who Achieved Disease Activity Index Score 28 Using C-reactive Protein (DAS28-CRP) Remission at Week 12
Description: Percentage of participants who achieved DAS28-CRP remission at Week 12 were reported. The DAS28 remission is defined as DAS28 -CRP value of less than (<) 2.6 at Week 12. The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity, and CRP; in mg/L). The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, MCP1 to MCP5, PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. Score on the DAS28 ranged from 0 to 10, where higher scores indicated more disease activity. Negative changes from baseline indicated improvement of arthritis.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Placebo | Group 2: Nipocalimab
Number analyzed (Participants) | 20 | 33
Percentage of Participants | 10.0 [-1.24 to 0.07] | 21.2 [-1.66 to -0.40]

7. Secondary Outcome: Percentage of Participants Who Achieved Disease Activity Index Score 28 Using C-reactive Protein (DAS28-CRP) Low Disease Activity (LDA) European League Against Rheumatism (EULAR) at Week 12
Description: Percentage of participants who achieved DAS28-CRP LDA EULAR at Week 12 were reported. The DAS28 LDA EULAR is defined as DAS28 -CRP value of less than or equal to (<=) 3.2 at Week 12. The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity, and C-reactive protein (CRP; in mg/L). The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, MCP1 to MCP5, PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. Score on the DAS28 ranged from 0 to 10, where higher scores indicated more disease activity. Negative changes from baseline indicated improvement of arthritis.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Placebo | Group 2: Nipocalimab
Number analyzed (Participants) | 20 | 33
Percentage of Participants | 10.0 [-1.24 to 0.07] | 21.2 [-1.66 to -0.40]

8. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score at Week 12
Description: Change from baseline in HAQ-DI score at Week 12 were reported. The HAQ-DI is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas: dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living, over the past week. Responses in each functional area were scored on a scale from 0 (indicating no difficulty) to 3 (inability to perform a task in that area). Overall score was computed as the sum of category scores and divided by the number of categories answered and ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability.
Time Frame: Baseline (Week 0), Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Group 1: Placebo | Group 2: Nipocalimab
Number analyzed (Participants) | 20 | 33
Score on a scale | -0.21 [-0.45 to 0.04] | -0.42 [-0.66 to -0.19]

9. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Percentage of participants with TEAEs were reported. An adverse event (AE) was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. TEAEs were defined as any AE occurring at or after the initial administration of study intervention through the safety follow-up visit (8 weeks after the last administration of study intervention).
Time Frame: From Week 0 up to 8 weeks post last dose at Week 10 (up to Week 18)
Population: The safety analysis set included all randomized participants who received at least 1 dose (partial or complete) of any study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Placebo | Group 2: Nipocalimab
Number analyzed (Participants) | 20 | 33
Percentage of Participants | 60.0 [-1.24 to 0.07] | 81.8 [-1.66 to -0.40]

10. Secondary Outcome: Percentage of Participants With Treatment-emergent Serious Adverse Events (TESAEs)
Description: Percentage of participants with TESAEs were reported. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. A SAE was any untoward medical occurrence at any dose that: resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/ incapacity, or resulted in congenital anomaly/birth defect. TESAEs were defined as any SAE occurring at or after the initial administration of study intervention through the safety follow-up visit (8 weeks after the last administration of study intervention).
Time Frame: From Week 0 up to 8 weeks post last dose at Week 10 (up to Week 18)
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Placebo | Group 2: Nipocalimab
Number analyzed (Participants) | 20 | 33
Percentage of Participants | 0 [-1.24 to 0.07] | 9.1 [-1.66 to -0.40]

11. Secondary Outcome: Percentage of Participants With AEs Leading to Discontinuation of Study Intervention
Description: Percentage of participants with AEs leading to discontinuation of study intervention were reported. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention.
Time Frame: From Week 0 up to Week 10
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Placebo | Group 2: Nipocalimab
Number analyzed (Participants) | 20 | 33
Percentage of Participants | 30.0 [-1.24 to 0.07] | 18.2 [-1.66 to -0.40]

12. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events of Special Interest (AESIs)
Description: Percentage of participants with TEAEs of special interest were reported. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. TEAEs were defined as any AE occurring at or after the initial administration of study intervention through the safety follow-up visit (8 weeks after the last administration of study intervention). TEAEs associated with the following situations were considered to be AESIs: (a) Infections that were severe or require IV anti-infective or operative/invasive intervention; (b) Hypoalbuminemia with albumin <20 grams per liter (g/L) (<2.0 grams per deciliter [g/dL]).
Time Frame: From Week 0 up to 8 weeks post last dose at Week 10 (up to Week 18)
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Placebo | Group 2: Nipocalimab
Number analyzed (Participants) | 20 | 33
Percentage of Participants | 0 [-1.24 to 0.07] | 3.0 [-1.66 to -0.40]

ADVERSE EVENTS:
Time Frame: All cause mortality: From screening (Week -6) up to Week 18; Serious and non-serious AEs: From Week 0 up to Week 18
Description: The safety analysis set included all randomized participants who received at least 1 dose (partial or complete) of any study intervention.
Arm/Group | Group 1: Placebo | Group 2: Nipocalimab
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/20 | 3/33
Other Adverse Events (participants affected / at risk) | 12/20 | 20/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Placebo (N=20) | Group 2: Nipocalimab (N=33)
Burn Infection (Infections and infestations) | 0 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Placebo (N=20) | Group 2: Nipocalimab (N=33)
Nausea (Gastrointestinal disorders) | 2 | 0
Paraesthesia Oral (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 2
Seasonal Allergy (Immune system disorders) | 1 | 0
Abscess Limb (Infections and infestations) | 1 | 0
Covid-19 (Infections and infestations) | 0 | 4
Cystitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2
Oral Herpes (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 2
Arthropod Bite (Injury, poisoning and procedural complications) | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0
Synovial Rupture (Injury, poisoning and procedural complications) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 9
Headache (Nervous system disorders) | 1 | 4
Nocturia (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT04991753/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT04991753/SAP_001.pdf